CLINICAL TRIAL: NCT03572972
Title: THE REAL WORLD EVIDENCE ON TREATMENT PATTERNS, EFFECTIVENESS, AND SAFETY OF DRUGS FOR STROKE PREVENTION IN NONVALVULAR ATRIAL FIBRILLATION PATIENTS IN KOREA
Brief Title: Non-interventional, Retrospective Cohort Study to Explore OAC Treatment in Korea
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: X9001134
Record Dates: First submitted 2018-06-19; First posted 2018-06-28 (Actual); Results first posted 2020-02-12 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2020-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — apixaban; Dabigatran; Rivaroxaban; Warfarin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (5):
- Patients prescribed apixaban
  Interventions: Drug: Apixaban
- Patients prescribed dabigatran
  Interventions: Drug: Dabigatran
- Patients prescribed rivaroxaban
  Interventions: Drug: Rivaroxaban
- Patients prescribed warfarin
  Interventions: Drug: warfarin
- Patients prescribed antiplatelet
  Interventions: Drug: Antiplatelets

INTERVENTIONS:
Drug: Apixaban — Treatment for NVAF patients
  Groups: Patients prescribed apixaban
Drug: Dabigatran — Treatment for NVAF patients
  Groups: Patients prescribed dabigatran
Drug: Rivaroxaban — Treatment for NVAF patients
  Groups: Patients prescribed rivaroxaban
Drug: warfarin — Treatment for NVAF patients
  Groups: Patients prescribed warfarin
Drug: Antiplatelets — Treatment for NVAF patients
  Groups: Patients prescribed antiplatelet

SUMMARY:
The primary purpose of this study is to evaluate comparative effectiveness and safety outcomes of therapies to prevent thromboembolic events in patients with nonvalvular atrial fibrillation by using Korean nationwide health claims database.

ELIGIBILITY:
Inclusion criteria:

1. Patients aged 18 years or older on the index date
2. Patients had ≥1 medical claim for AF (refer to Table 1) before or on the index date with at least one hospitalization or at least two outpatient visits:
3. Patients prescribed aspirin, warfarin, or NOACs during intake period (from July 1, 2015 to November 30, 2016)

Exclusion criteria:

Patients meeting any of the following criteria will not be included in the study.

1. Medical claims indicating diagnosis or procedure for hip/knee replacement surgery within 6 weeks prior to index date
2. Medical claims indicating a diagnosis code indicative of rheumatic mitral valvular heart disease, mitral valve stenosis during the 12-month baseline period (Valvular AF / Prosthetic heart valves)
3. Medical claims indicating a diagnosis code of VTE (Venous thromboembolism) during the 12-month baseline period
4. Medical claims indicating a diagnosis or procedure code of transient AF, or cardiac surgery during the 12-month baseline period (Thyrotoxicosis, Hypertrophic cardiomyopathy, Elective defibrillation, radiofrequency ablation, or left atrial appendage occlusion)
5. Medical claims indicating a diagnosis code of other conditions during the 12-month baseline period (End-stage chronic kidney disease / Kidney transplant / Dialysis / Pericarditis)
6. For the comparison of "NOAC versus NOAC", and "NOAC versus warfarin", patients with any OACs (apixaban, dabigatran, rivaroxaban, or warfarin) in the pre-index period (from 1 year prior to the day before index date)
7. For the comparison of "NOAC versus aspirin", patients with following medications in the pre-index period (from 1 year prior to the day before index date)

   * NOAC user: OACs (apixaban, dabigatran, rivaroxaban, warfarin)
   * Aspirin user: none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from Korean Health Insurance Review & Assessment Service (HIRA) database according to the inclusion/exclusion criteria. Only users of oral anticoagulant or antiplatelet treatment for atrial fibrillation from July 1, 2015 to November 30, 2016 will be included in this study.
Sampling Method: Probability Sample
Enrollment: 64684 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Korea University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Lee MY, Han S, Bang OY, On YK, Jang SW, Han S, Ryu J, Park YJ, Kang S, Suh HS, Kim YH. Drug Utilization Pattern of Oral Anticoagulants in Patients with Atrial Fibrillation: A Nationwide Population-Based Study in Korea. Adv Ther. 2022 Jul;39(7):3112-3130. doi: 10.1007/s12325-022-02151-z. Epub 2022 May 7. PMID 35524839
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=X9001134

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data was retrieved from Korean Health Insurance Review & Assessment Service (HIRA) database, of participants who were diagnosed with non-valvular atrial fibrillation (NVAF) from 1-January-2007 up to and including index date, who newly initiated non-vitamin K antagonist oral anticoagulants (NOACs), warfarin or used aspirin during intake duration.
Pre-assignment Details: It is a retrospective, observational study. Index date: first prescription date of study drugs during intake duration. Intake period: between 1-July-2015 to 30-November-2016. Inverse probability of treatment weighted (IPTW) method was used to analyze outcome measures to balance participant's characteristics among reporting arms.
Groups:
- NOAC - Apixaban: Oral anticoagulants (OACs) treatment-naive participants diagnosed with NVAF, who initiated apixaban on the index date, were included in this study cohort and their data available in Korean HIRA database was retrospectively observed. Index date for apixaban was defined as the first prescription date of apixaban during the intake period from 1-July-2015 to 30-November-2016.
- NOAC - Dabigatran: OACs treatment-naive participants diagnosed with NVAF, who initiated dabigatran on the index date, were included in this study cohort and their data available in Korean HIRA database was retrospectively observed. Index date for dabigatran was defined as the first prescription date of dabigatran during the intake period from 1-July-2015 to 30-November-2016.
- NOAC - Rivaroxaban: OACs treatment-naive participants diagnosed with NVAF, who initiated rivaroxaban on the index date, were included in this study cohort and their data available in Korean HIRA database was retrospectively observed. Index date for rivaroxaban was defined as the first prescription date of rivaroxaban during the intake period from 1-July-2015 to 30-November-2016.
- Warfarin: OACs treatment-naive participants diagnosed with NVAF, who initiated warfarin on the index date, were included in this study cohort and their data available in Korean HIRA database was retrospectively observed. Index date for warfarin was defined as the first prescription date of warfarin during the intake period from 1-July-2015 to 30-November-2016.
- Aspirin: OACs treatment-naive participants diagnosed with NVAF, who initiated aspirin on the index date, were included in this study cohort and their data available in Korean HIRA database was retrospectively observed. Index date for aspirin was defined as the first prescription date of aspirin during the intake period from 1-July-2015 to 30-November-2016.
Period: Overall Study
Arm/Group | NOAC - Apixaban | NOAC - Dabigatran | NOAC - Rivaroxaban | Warfarin | Aspirin
Started | 10548 | 11414 | 17779 | 8648 | 16295
Completed | 10548 | 11414 | 17779 | 8648 | 16295
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: OACs treatment-naive participants diagnosed with NVAF, initiating warfarin, NOACs (apixaban, dabigatran, rivaroxaban) or aspirin treatment from 1-July-2015 to 30-November-2016.
Groups:
- Total: Total of all reporting groups
Arm/Group | NOAC - Apixaban | NOAC - Dabigatran | NOAC - Rivaroxaban | Warfarin | Aspirin | Total
Number analyzed (Participants) | 10548 | 11414 | 17779 | 8648 | 16295 | 64684
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.89 (9.52) | 72.23 (9.52) | 73.27 (9.55) | 68.73 (12.62) | 72.10 (9.17) | 72.29 (10.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5148 | 4926 | 8169 | 3238 | 6995 | 28476
  Male | 5400 | 6488 | 9610 | 5410 | 9300 | 36208
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Event Rate of Stroke/Systemic Embolism Requiring Hospitalization: NOAC Versus Warfarin Analysis
Description: Event rate was defined as number of events divided by 100 participant-years. Hemorrhagic stroke, ischemic stroke and systemic embolism requiring hospitalization identified using hospital claims which had hemorrhagic, ischemic stroke or systemic embolism Korean standard classification of diseases (KCD) code, whichever came first (first occurred event used). KCD code: hemorrhagic stroke = I60-62, I690-692; ischemic stroke = G459, I63, I693; systemic embolism = I74. Hospitalization and brain CT/MRI codes were used for ischemic stroke, hemorrhagic stroke.Hospitalization and any CT/MRI codes were used for systemic embolism. Index date = the first prescription date of study drugs during intake duration. Participants were identified as NOAC user or Warfarin user depending on the date when they first used NOAC or Warfarin during intake duration.
Time Frame: Maximum of 1 year 4 months (From 1-July-2015 to 30-November-2016)
Population: OACs treatment-naive participants with NVAF, starting any OACs in intake duration; matched on propensity scores by IPTW method to balance participant characteristics among specified arms. It created virtual groups used in analysis here. No data for Aspirin arm: could not be matched using IPTW with other arms due to heterogeneity characteristics.
Measure: Number; unit: events per 100 participants-years
Groups:
- Apixaban vs Warfarin (Apixaban): OACs treatment-naive participants diagnosed with NVAF, with index treatment of apixaban and matched on propensity scores with warfarin using inverse probability of treatment weighting (IPTW).
- Apixaban vs Warfarin (Warfarin): OACs treatment-naive participants diagnosed with NVAF, with index treatment of warfarin and matched on propensity scores with apixaban using IPTW.
- Dabigatran vs Warfarin (Dabigatran): OACs treatment-naive participants diagnosed with NVAF, with index treatment of dabigatran and matched on propensity scores with warfarin using IPTW.
- Dabigatran vs Warfarin (Warfarin): OACs treatment-naive participants diagnosed with NVAF, with index treatment of warfarin and matched on propensity scores with dabigatran using IPTW.
- Rivaroxaban vs Warfarin (Rivaroxaban): OACs treatment-naive participants diagnosed with NVAF, with index treatment of rivaroxaban and matched on propensity scores with warfarin using IPTW.
- Rivaroxaban vs Warfarin (Warfarin): OACs treatment-naive participants diagnosed with NVAF, with index treatment of warfarin and matched on propensity scores with rivaroxaban using IPTW.
Arm/Group | Apixaban vs Warfarin (Apixaban) | Apixaban vs Warfarin (Warfarin) | Dabigatran vs Warfarin (Dabigatran) | Dabigatran vs Warfarin (Warfarin) | Rivaroxaban vs Warfarin (Rivaroxaban) | Rivaroxaban vs Warfarin (Warfarin)
Number analyzed (Participants) | 10514 | 8677 | 11415 | 8676 | 17780 | 8638
events per 100 participants-years | 7.66 | 13.52 | 7.2 | 13.53 | 7.18 | 12.89
Statistical Analysis 1: Comparison: Apixaban vs Warfarin (Apixaban) vs Apixaban vs Warfarin (Warfarin); Cox proportional hazards model was used to compare event rates between the treatment groups. To check the proportional hazards assumption, the graphical methods and statistical tests using the time-dependent covariate were used. If there were evidence of violation in the proportional hazards assumption in graphical methods, the statistical tests were used and if the evidence of assumption violation still existed, the value of hazard ratio (HR) at year 1 as an extended Cox model was used; Test type: Superiority; Hazard Ratio (HR) = 0.618, 95% CI 2-sided [0.541 to 0.707]
Statistical Analysis 2: Comparison: Dabigatran vs Warfarin (Dabigatran) vs Dabigatran vs Warfarin (Warfarin); Cox proportional hazards model was used to compare event rates between the treatment groups. To check the proportional hazards assumption, the graphical methods and statistical tests using the time-dependent covariate were used. If there were evidence of violation in the proportional hazards assumption in graphical methods, the statistical tests were used and if the evidence of assumption violation still existed, the value of HR at year 1 as an extended Cox model was used; Test type: Superiority; Hazard Ratio (HR) = 0.604, 95% CI 2-sided [0.530 to 0.687]
Statistical Analysis 3: Comparison: Rivaroxaban vs Warfarin (Rivaroxaban) vs Rivaroxaban vs Warfarin (Warfarin); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.705, 95% CI 2-sided [0.563 to 0.884] — HR evaluated using extended Cox model

2. Primary Outcome: Event Rate of Stroke/Systemic Embolism Requiring Hospitalization: NOAC Versus NOAC Analysis
Description: Event rate was defined as number of events divided by 100 participant-years. Hemorrhagic stroke, ischemic stroke and systemic embolism requiring hospitalization identified using hospital claims which had hemorrhagic, ischemic stroke or systemic embolism Korean standard classification of diseases (KCD) code, whichever came first (first occurred event used). KCD code: hemorrhagic stroke = I60-62, I690-692; ischemic stroke = G459, I63, I693; systemic embolism = I74. Hospitalization and brain CT/MRI codes were used for ischemic stroke, hemorrhagic stroke.Hospitalization and any CT/MRI codes were used for systemic embolism. Index date = the first prescription date of study drugs during intake duration.
Time Frame: Maximum of 1 year 4 months (From 1-July-2015 to 30-November-2016)
Population: as for outcome 1
Measure: Number; unit: events per 100 participants-years
Groups:
- Apixaban vs Dabigatran (Apixaban): OACs treatment-naive participants diagnosed with NVAF, with index treatment of apixaban and matched on propensity scores with dabigatran using IPTW.
- Apixaban vs Dabigatran (Dabigatran): OACs treatment-naive participants diagnosed with NVAF, with index treatment of dabigatran and matched on propensity scores with apixaban using IPTW.
- Apixaban vs Rivaroxaban (Apixaban): OACs treatment-naive participants diagnosed with NVAF, with index treatment of apixaban and matched on propensity scores with rivaroxaban using IPTW.
- Apixaban vs Rivaroxaban (Rivaroxaban): OACs treatment-naive participants diagnosed with NVAF, with index treatment of rivaroxaban and matched on propensity scores with apixaban using IPTW.
- Dabigatran vs Rivaroxaban (Dabigatran): OACs treatment-naive participants diagnosed with NVAF, with index treatment of dabigatran and matched on propensity scores with rivaroxaban using IPTW.
- Dabigatran vs Rivaroxaban (Rivaroxaban): OACs treatment-naive participants diagnosed with NVAF, with index treatment of rivaroxaban and matched on propensity scores with dabigatran using IPTW.
Arm/Group | Apixaban vs Dabigatran (Apixaban) | Apixaban vs Dabigatran (Dabigatran) | Apixaban vs Rivaroxaban (Apixaban) | Apixaban vs Rivaroxaban (Rivaroxaban) | Dabigatran vs Rivaroxaban (Dabigatran) | Dabigatran vs Rivaroxaban (Rivaroxaban)
Number analyzed (Participants) | 10567 | 11415 | 10545 | 17812 | 11416 | 17801
events per 100 participants-years | 7.75 | 7.47 | 7.35 | 7.48 | 7.01 | 7.31
Statistical Analysis 1: Comparison: Apixaban vs Dabigatran (Apixaban) vs Apixaban vs Dabigatran (Dabigatran); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.993, 95% CI 2-sided [0.870 to 1.134]
Statistical Analysis 2: Comparison: Apixaban vs Rivaroxaban (Apixaban) vs Apixaban vs Rivaroxaban (Rivaroxaban); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.949, 95% CI 2-sided [0.839 to 1.073]
Statistical Analysis 3: Comparison: Dabigatran vs Rivaroxaban (Dabigatran) vs Dabigatran vs Rivaroxaban (Rivaroxaban); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.961, 95% CI 2-sided [0.854 to 1.082]

3. Primary Outcome: Event Rate of Major Bleeding Requiring Hospitalization: NOAC Versus Warfarin Analysis
Description: Event rate: number of events divided by 100 participant-years. Intracranial hemorrhage (ICH), gastrointestinal (GI) bleeding and other bleeding requiring hospitalization identified using hospital claims which had ICH, GI and other bleeding KCD code whichever came first (first occurred event used). KCD code: ICH = I60-62, I690-92, S064-66, S068; GI bleeding = I850, I983, K2211, K226, K228, K250, K252, K254, K256, K260, K262, K264, K266, K270, K272, K274, K276, K280, K282, K284, K286, K290, K3181, K5521, K625, K920, K921, K922; other bleeding = D62,H448,H3572,H356,H313,H210,H113,H052,H470,H431,I312,N020-N029,N421,N831,N857,N920,N923,N930,N938-939,M250,R233,R040-042,R048-049,T792,T810,N950,R310, R311, R318, R58, T455, Y442, D683). Brain CT/MRI codes were used for ICH only. Index date= first prescription date of study drugs during intake duration. Participants were identified as NOAC user/Warfarin user depending on the date when they first used NOAC or Warfarin during intake duration.
Time Frame: Maximum of 1 year 4 months (From 1-July-2015 to 30-November-2016)
Population: as for outcome 1
Measure: Number; unit: events per 100 participants-years
Groups:
- Apixaban vs Warfarin (Apixaban): OACs treatment-naive participants diagnosed with NVAF, with index treatment of apixaban and matched on propensity scores with warfarin using IPTW.
Arm/Group | Apixaban vs Warfarin (Apixaban) | Apixaban vs Warfarin (Warfarin) | Dabigatran vs Warfarin (Dabigatran) | Dabigatran vs Warfarin (Warfarin) | Rivaroxaban vs Warfarin (Rivaroxaban) | Rivaroxaban vs Warfarin (Warfarin)
Number analyzed (Participants) | 10514 | 8677 | 11415 | 8676 | 17780 | 8638
events per 100 participants-years | 7.97 | 14.73 | 8.57 | 13.77 | 9.55 | 14.23
Statistical Analysis 1: Comparison: Apixaban vs Warfarin (Apixaban) vs Apixaban vs Warfarin (Warfarin); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.583, 95% CI 2-sided [0.512 to 0.664]
Statistical Analysis 2: Comparison: Dabigatran vs Warfarin (Dabigatran) vs Dabigatran vs Warfarin (Warfarin); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.754, 95% CI 2-sided [0.597 to 0.953] — HR evaluated using extended Cox model
Statistical Analysis 3: Comparison: Rivaroxaban vs Warfarin (Rivaroxaban) vs Rivaroxaban vs Warfarin (Warfarin); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.844, 95% CI 2-sided [0.685 to 1.040] — HR evaluated using extended Cox model

4. Primary Outcome: Event Rate of Major Bleeding Requiring Hospitalization: NOAC Versus NOAC Analysis
Description: Event rate was defined as number of events divided by 100 participant-years. Intracranial hemorrhage (ICH), gastrointestinal (GI) bleeding and other bleeding requiring hospitalization identified using hospital claims which had ICH, GI and other bleeding KCD code whichever came first (first occurred event used). KCD code: ICH = I60-62, I690-92, S064-66, S068; GI bleeding = I850, I983, K2211, K226, K228, K250, K252, K254, K256, K260, K262, K264, K266, K270, K272, K274, K276, K280, K282, K284, K286, K290, K3181, K5521, K625, K920, K921, K922; other bleeding = D62, H448, H3572, H356, H313, H210, H113, H052, H470, H431, I312, N020-N029, N421, N831, N857, N920, N923, N930, N938-939, M250, R233, R040-042, R048-049, T792, T810, N950, R310, R311, R318, R58, T455, Y442, D683). Brain CT/MRI codes were used for ICH only. Index date = the first prescription date of study drugs during intake duration.
Time Frame: Maximum of 1 year 4 months (From 1-July-2015 to 30-November-2016)
Population: as for outcome 1
Measure: Number; unit: events per 100 participants-years
Arm/Group | Apixaban vs Dabigatran (Apixaban) | Apixaban vs Dabigatran (Dabigatran) | Apixaban vs Rivaroxaban (Apixaban) | Apixaban vs Rivaroxaban (Rivaroxaban) | Dabigatran vs Rivaroxaban (Dabigatran) | Dabigatran vs Rivaroxaban (Rivaroxaban)
Number analyzed (Participants) | 10567 | 11415 | 10545 | 17812 | 11416 | 17801
events per 100 participants-years | 7.70 | 8.65 | 7.77 | 9.86 | 8.18 | 9.36
Statistical Analysis 1: Comparison: Apixaban vs Dabigatran (Apixaban) vs Apixaban vs Dabigatran (Dabigatran); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.866, 95% CI 2-sided [0.761 to 0.985]
Statistical Analysis 2: Comparison: Apixaban vs Rivaroxaban (Apixaban) vs Apixaban vs Rivaroxaban (Rivaroxaban); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.768, 95% CI 2-sided [0.684 to 0.862]
Statistical Analysis 3: Comparison: Dabigatran vs Rivaroxaban (Dabigatran) vs Dabigatran vs Rivaroxaban (Rivaroxaban); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.875, 95% CI 2-sided [0.786 to 0.975]

5. Secondary Outcome: Event Rate of Hemorrhagic Stroke Requiring Hospitalization: NOAC Versus Warfarin Analysis
Description: Event rate was number of events divided by 100 participant-years for first occurrence of hemorrhagic stroke events after index date was reported. Hemorrhagic stroke requiring hospitalization was identified using hospital claims which had a hemorrhagic stroke KCD code (I60-62, I690-692). For hemorrhagic stroke, hospitalization and brain CT or MRI codes were also required. Index date = the first prescription date of study drugs during intake duration. Participants were identified as NOAC user or Warfarin user depending on the date when they first used NOAC or Warfarin during intake duration.
Time Frame: Maximum of 1 year 4 months (From 1-July-2015 to 30-November-2016)
Population: as for outcome 1
Measure: Number; unit: events per 100 participants-years
Arm/Group | Apixaban vs Warfarin (Apixaban) | Apixaban vs Warfarin (Warfarin) | Dabigatran vs Warfarin (Dabigatran) | Dabigatran vs Warfarin (Warfarin) | Rivaroxaban vs Warfarin (Rivaroxaban) | Rivaroxaban vs Warfarin (Warfarin)
Number analyzed (Participants) | 10514 | 8677 | 11415 | 8676 | 17780 | 8638
events per 100 participants-years | 1.1 | 1.73 | 0.78 | 1.71 | 1.18 | 1.72
Statistical Analysis 1: Comparison: Apixaban vs Warfarin (Apixaban) vs Apixaban vs Warfarin (Warfarin); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.673, 95% CI 2-sided [0.470 to 0.964]
Statistical Analysis 2: Comparison: Dabigatran vs Warfarin (Dabigatran) vs Dabigatran vs Warfarin (Warfarin); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.491, 95% CI 2-sided [0.337 to 0.715]
Statistical Analysis 3: Comparison: Rivaroxaban vs Warfarin (Rivaroxaban) vs Rivaroxaban vs Warfarin (Warfarin); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.747, 95% CI 2-sided [0.548 to 1.018]

6. Secondary Outcome: Event Rate of Hemorrhagic Stroke Requiring Hospitalization: NOAC Versus NOAC Analysis
Description: Event rate was defined as number of events divided by 100 participant-years for first occurrence of hemorrhagic stroke events after index date was reported. Hemorrhagic stroke requiring hospitalization was identified using hospital claims which had a hemorrhagic stroke KCD code (I60-62, I690-692). For hemorrhagic stroke, hospitalization and brain CT or MRI codes were also required. Index date = the first prescription date of study drugs during intake duration.
Time Frame: Maximum of 1 year 4 months (From 1-July-2015 to 30-November-2016)
Population: as for outcome 1
Measure: Number; unit: events per 100 participants-years
Arm/Group | Apixaban vs Dabigatran (Apixaban) | Apixaban vs Dabigatran (Dabigatran) | Apixaban vs Rivaroxaban (Apixaban) | Apixaban vs Rivaroxaban (Rivaroxaban) | Dabigatran vs Rivaroxaban (Dabigatran) | Dabigatran vs Rivaroxaban (Rivaroxaban)
Number analyzed (Participants) | 10567 | 11415 | 10545 | 17812 | 11416 | 17801
events per 100 participants-years | 1.11 | 0.74 | 1.05 | 1.15 | 0.71 | 1.14
Statistical Analysis 1: Comparison: Apixaban vs Dabigatran (Apixaban) vs Apixaban vs Dabigatran (Dabigatran); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 1.463, 95% CI 2-sided [0.998 to 2.145]
Statistical Analysis 2: Comparison: Apixaban vs Rivaroxaban (Apixaban) vs Apixaban vs Rivaroxaban (Rivaroxaban); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.890, 95% CI 2-sided [0.647 to 1.225]
Statistical Analysis 3: Comparison: Dabigatran vs Rivaroxaban (Dabigatran) vs Dabigatran vs Rivaroxaban (Rivaroxaban); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.630, 95% CI 2-sided [0.447 to 0.888]

7. Secondary Outcome: Event Rate of Ischemic Stroke Requiring Hospitalization: NOAC Versus Warfarin Analysis
Description: Event rate was defined as number of events divided by 100 participant-years for first occurrence of ischemic stroke events after index date was reported. Ischemic stroke requiring hospitalization was identified using hospital claims which had ischemic stroke KCD code (G459, I63, and I693). For ischemic stroke, hospitalization and brain CT or MRI codes were also required. Index date = the first prescription date of study drugs during intake duration. Participants were identified as NOAC user or Warfarin user depending on the date when they first used NOAC or Warfarin during intake duration.
Time Frame: Maximum of 1 year 4 months (From 1-July-2015 to 30-November-2016)
Population: as for outcome 1
Measure: Number; unit: events per 100 participants-years
Arm/Group | Apixaban vs Warfarin (Apixaban) | Apixaban vs Warfarin (Warfarin) | Dabigatran vs Warfarin (Dabigatran) | Dabigatran vs Warfarin (Warfarin) | Rivaroxaban vs Warfarin (Rivaroxaban) | Rivaroxaban vs Warfarin (Warfarin)
Number analyzed (Participants) | 10514 | 8677 | 11415 | 8676 | 17780 | 8638
events per 100 participants-years | 6.9 | 11.8 | 6.53 | 11.92 | 6.29 | 11.19
Statistical Analysis 1: Comparison: Apixaban vs Warfarin (Apixaban) vs Apixaban vs Warfarin (Warfarin); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.640, 95% CI 2-sided [0.556 to 0.738]
Statistical Analysis 2: Comparison: Dabigatran vs Warfarin (Dabigatran) vs Dabigatran vs Warfarin (Warfarin); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.624, 95% CI 2-sided [0.544 to 0.715]
Statistical Analysis 3: Comparison: Rivaroxaban vs Warfarin (Rivaroxaban) vs Rivaroxaban vs Warfarin (Warfarin); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.749, 95% CI 2-sided [0.588 to 0.954] — HR evaluated using extended Cox model

8. Secondary Outcome: Event Rate of Ischemic Stroke Requiring Hospitalization: NOAC Versus NOAC Analysis
Description: Event rate was defined as number of events divided by 100 participant-years for first occurrence of ischemic stroke events after index date was reported. Ischemic stroke requiring hospitalization was identified using hospital claims which had ischemic stroke KCD code (G459, I63, and I693). For ischemic stroke, hospitalization and brain CT or MRI codes were also required. Index date = the first prescription date of study drugs during intake duration.
Time Frame: Maximum of 1 year 4 months (From 1-July-2015 to 30-November-2016)
Population: as for outcome 1
Measure: Number; unit: events per 100 participants-years
Arm/Group | Apixaban vs Dabigatran (Apixaban) | Apixaban vs Dabigatran (Dabigatran) | Apixaban vs Rivaroxaban (Apixaban) | Apixaban vs Rivaroxaban (Rivaroxaban) | Dabigatran vs Rivaroxaban (Dabigatran) | Dabigatran vs Rivaroxaban (Rivaroxaban)
Number analyzed (Participants) | 10567 | 11415 | 10545 | 17812 | 11416 | 17801
events per 100 participants-years | 6.99 | 6.84 | 6.60 | 6.58 | 6.37 | 6.43
Statistical Analysis 1: Comparison: Apixaban vs Dabigatran (Apixaban) vs Apixaban vs Dabigatran (Dabigatran); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.977, 95% CI 2-sided [0.850 to 1.122]
Statistical Analysis 2: Comparison: Apixaban vs Rivaroxaban (Apixaban) vs Apixaban vs Rivaroxaban (Rivaroxaban); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.966, 95% CI 2-sided [0.848 to 1.100]
Statistical Analysis 3: Comparison: Dabigatran vs Rivaroxaban (Dabigatran) vs Dabigatran vs Rivaroxaban (Rivaroxaban); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.993, 95% CI 2-sided [0.877 to 1.125]

9. Secondary Outcome: Event Rate of Systemic Embolism Requiring Hospitalization: NOAC Versus Warfarin Analysis
Description: Event rate was defined as number of events divided by 100 participant-years for first occurrence of systemic embolism. Systemic embolism requiring hospitalization was identified using hospital claims which had systemic embolism KCD code = I74. For systemic embolism, hospitalization and any CT or MRI codes was used. Index date = the first prescription date of study drugs during intake duration. Participants were identified as NOAC user or Warfarin user depending on the date when they first used NOAC or Warfarin during intake duration
Time Frame: Maximum of 1 year 4 months (From 1-July-2015 to 30-November-2016)
Population: as for outcome 1
Measure: Number; unit: events per 100 participants-years
Arm/Group | Apixaban vs Warfarin (Apixaban) | Apixaban vs Warfarin (Warfarin) | Dabigatran vs Warfarin (Dabigatran) | Dabigatran vs Warfarin (Warfarin) | Rivaroxaban vs Warfarin (Rivaroxaban) | Rivaroxaban vs Warfarin (Warfarin)
Number analyzed (Participants) | 10514 | 8677 | 11415 | 8676 | 17780 | 8638
events per 100 participants-years | 0.18 | 0.78 | 0.24 | 0.75 | 0.27 | 0.74
Statistical Analysis 1: Comparison: Apixaban vs Warfarin (Apixaban) vs Apixaban vs Warfarin (Warfarin); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.250, 95% CI 2-sided [0.119 to 0.523]
Statistical Analysis 2: Comparison: Dabigatran vs Warfarin (Dabigatran) vs Dabigatran vs Warfarin (Warfarin); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.380, 95% CI 2-sided [0.203 to 0.711]
Statistical Analysis 3: Comparison: Rivaroxaban vs Warfarin (Rivaroxaban) vs Rivaroxaban vs Warfarin (Warfarin); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.422, 95% CI 2-sided [0.247 to 0.722]

10. Secondary Outcome: Event Rate of Systemic Embolism Requiring Hospitalization: NOAC Versus NOAC Analysis
Description: Event rate was defined as number of events divided by 100 participant-years for first occurrence of systemic embolism. Systemic embolism requiring hospitalization was identified using hospital claims which had systemic embolism KCD code = I74. For systemic embolism, hospitalization and any CT or MRI codes was used. Index date= the first prescription date of study drugs during intake duration.
Time Frame: Maximum of 1 year 4 months (From 1-July-2015 to 30-November-2016)
Population: as for outcome 1
Measure: Number; unit: events per 100 participants-years
Arm/Group | Apixaban vs Dabigatran (Apixaban) | Apixaban vs Dabigatran (Dabigatran) | Apixaban vs Rivaroxaban (Apixaban) | Apixaban vs Rivaroxaban (Rivaroxaban) | Dabigatran vs Rivaroxaban (Dabigatran) | Dabigatran vs Rivaroxaban (Rivaroxaban)
Number analyzed (Participants) | 10567 | 11415 | 10545 | 17812 | 11416 | 17801
events per 100 participants-years | 0.20 | 0.25 | 0.20 | 0.28 | 0.24 | 0.26
Statistical Analysis 1: Comparison: Apixaban vs Dabigatran (Apixaban) vs Apixaban vs Dabigatran (Dabigatran); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.745, 95% CI 2-sided [0.343 to 1.615]
Statistical Analysis 2: Comparison: Apixaban vs Rivaroxaban (Apixaban) vs Apixaban vs Rivaroxaban (Rivaroxaban); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.692, 95% CI 2-sided [0.342 to 1.402]
Statistical Analysis 3: Comparison: Dabigatran vs Rivaroxaban (Dabigatran) vs Dabigatran vs Rivaroxaban (Rivaroxaban); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.932, 95% CI 2-sided [0.498 to 1.747]

11. Secondary Outcome: Event Rate of Gastrointestinal (GI) Bleeding Requiring Hospitalization: NOAC Versus Warfarin Analysis
Description: Event rate was defined as number of events divided by 100 participant-years for first occurrence of GI bleeding events after index date was reported. GI bleeding requiring hospitalization was identified using hospital claims which had a GI bleeding KCD code (I850, I983, K2211, K226, K228, K250, K252, K254, K256, K260, K262, K264, K266, K270, K272, K274, K276, K280, K282, K284, K286, K290, K3181, K5521, K625, K920, K921, K922). Index date = the first prescription date of study drugs during intake duration. Participants were identified as NOAC user or Warfarin user depending on the date when they first used NOAC or Warfarin during intake duration.
Time Frame: Maximum of 1 year 4 months (From 1-July-2015 to 30-November-2016)
Population: as for outcome 1
Measure: Number; unit: events per 100 participants-years
Arm/Group | Apixaban vs Warfarin (Apixaban) | Apixaban vs Warfarin (Warfarin) | Dabigatran vs Warfarin (Dabigatran) | Dabigatran vs Warfarin (Warfarin) | Rivaroxaban vs Warfarin (Rivaroxaban) | Rivaroxaban vs Warfarin (Warfarin)
Number analyzed (Participants) | 10514 | 8677 | 11415 | 8676 | 17780 | 8638
events per 100 participants-years | 3.44 | 6.2 | 4.17 | 5.56 | 4.32 | 5.78
Statistical Analysis 1: Comparison: Apixaban vs Warfarin (Apixaban) vs Apixaban vs Warfarin (Warfarin); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.600, 95% CI 2-sided [0.492 to 0.731]
Statistical Analysis 2: Comparison: Dabigatran vs Warfarin (Dabigatran) vs Dabigatran vs Warfarin (Warfarin); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 1.046, 95% CI 2-sided [0.719 to 1.522] — HR evaluated using extended Cox model
Statistical Analysis 3: Comparison: Rivaroxaban vs Warfarin (Rivaroxaban) vs Rivaroxaban vs Warfarin (Warfarin); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 1.295, 95% CI 2-sided [0.920 to 1.824] — HR evaluated using extended Cox model

12. Secondary Outcome: Event Rate of Gastrointestinal (GI) Bleeding Requiring Hospitalization: NOAC Versus NOAC Analysis
Description: Event rate was defined as number of events divided by 100 participant-years for first occurrence of GI bleeding events after index date was reported. GI bleeding requiring hospitalization was identified using hospital claims which had a GI bleeding KCD code (I850, I983, K2211, K226, K228, K250, K252, K254, K256, K260, K262, K264, K266, K270, K272, K274, K276, K280, K282, K284, K286, K290, K3181, K5521, K625, K920, K921, K922). Index date = the first prescription date of study drugs during intake duration.
Time Frame: Maximum of 1 year 4 months (From 1-July-2015 to 30-November-2016)
Population: as for outcome 1
Measure: Number; unit: events per 100 participants-years
Arm/Group | Apixaban vs Dabigatran (Apixaban) | Apixaban vs Dabigatran (Dabigatran) | Apixaban vs Rivaroxaban (Apixaban) | Apixaban vs Rivaroxaban (Rivaroxaban) | Dabigatran vs Rivaroxaban (Dabigatran) | Dabigatran vs Rivaroxaban (Rivaroxaban)
Number analyzed (Participants) | 10567 | 11415 | 10545 | 17812 | 11416 | 17801
events per 100 participants-years | 3.23 | 4.18 | 3.28 | 4.59 | 3.97 | 4.25
Statistical Analysis 1: Comparison: Apixaban vs Dabigatran (Apixaban) vs Apixaban vs Dabigatran (Dabigatran); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.751, 95% CI 2-sided [0.62 to 0.91]
Statistical Analysis 2: Comparison: Apixaban vs Rivaroxaban (Apixaban) vs Apixaban vs Rivaroxaban (Rivaroxaban); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.697, 95% CI 2-sided [0.586 to 0.830]
Statistical Analysis 3: Comparison: Dabigatran vs Rivaroxaban (Dabigatran) vs Dabigatran vs Rivaroxaban (Rivaroxaban); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.936, 95% CI 2-sided [0.801 to 1.094]

13. Secondary Outcome: Event Rate of Intracranial Hemorrhage Requiring Hospitalization: NOAC Versus Warfarin Analysis
Description: Event rate was defined as number of events divided by 100 participant-years for first occurrence of intracranial hemorrhage events after index date was reported. Intracranial hemorrhage requiring hospitalization was identified using hospital claims which had an intracranial hemorrhage KCD code (I60, I61, I62, I690, I691, I692, S064, S065, S066, and S068) and brain CT or MRI codes. Index date = the first prescription date of study drugs during intake duration. Participants were identified as NOAC user or Warfarin user depending on the date when they first used NOAC or Warfarin during intake duration.
Time Frame: Maximum of 1 year 4 months (From 1-July-2015 to 30-November-2016)
Population: as for outcome 1
Measure: Number; unit: events per 100 participants-years
Arm/Group | Apixaban vs Warfarin (Apixaban) | Apixaban vs Warfarin (Warfarin) | Dabigatran vs Warfarin (Dabigatran) | Dabigatran vs Warfarin (Warfarin) | Rivaroxaban vs Warfarin (Rivaroxaban) | Rivaroxaban vs Warfarin (Warfarin)
Number analyzed (Participants) | 10514 | 8677 | 11415 | 8676 | 17780 | 8638
events per 100 participants-years | 1.37 | 2.38 | 1.17 | 2.31 | 1.47 | 2.37
Statistical Analysis 1: Comparison: Apixaban vs Warfarin (Apixaban) vs Apixaban vs Warfarin (Warfarin); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.373, 95% CI 2-sided [0.212 to 0.658] — HR evaluated using extended Cox model
Statistical Analysis 2: Comparison: Dabigatran vs Warfarin (Dabigatran) vs Dabigatran vs Warfarin (Warfarin); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.538, 95% CI 2-sided [0.392 to 0.737]
Statistical Analysis 3: Comparison: Rivaroxaban vs Warfarin (Rivaroxaban) vs Rivaroxaban vs Warfarin (Warfarin); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.664, 95% CI 2-sided [0.507 to 0.870]

14. Secondary Outcome: Event Rate of Intracranial Hemorrhage Requiring Hospitalization: NOAC Versus NOAC Analysis
Description: Event rate was defined as number of events divided by 100 participant-years for first occurrence of intracranial hemorrhage events after index date was reported. Intracranial hemorrhage requiring hospitalization was identified using hospital claims which had an intracranial hemorrhage KCD code (I60, I61, I62, I690, I691, I692, S064, S065, S066, and S068) and brain CT or MRI codes. Index date = the first prescription date of study drugs during intake duration.
Time Frame: Maximum of 1 year 4 months (From 1-July-2015 to 30-November-2016)
Population: as for outcome 1
Measure: Number; unit: events per 100 participants-years
Arm/Group | Apixaban vs Dabigatran (Apixaban) | Apixaban vs Dabigatran (Dabigatran) | Apixaban vs Rivaroxaban (Apixaban) | Apixaban vs Rivaroxaban (Rivaroxaban) | Dabigatran vs Rivaroxaban (Dabigatran) | Dabigatran vs Rivaroxaban (Rivaroxaban)
Number analyzed (Participants) | 10567 | 11415 | 10545 | 17812 | 11416 | 17801
events per 100 participants-years | 1.39 | 1.12 | 1.35 | 1.43 | 1.08 | 1.41
Statistical Analysis 1: Comparison: Apixaban vs Dabigatran (Apixaban) vs Apixaban vs Dabigatran (Dabigatran); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 1.204, 95% CI 2-sided [0.871 to 1.666]
Statistical Analysis 2: Comparison: Apixaban vs Rivaroxaban (Apixaban) vs Apixaban vs Rivaroxaban (Rivaroxaban); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.918, 95% CI 2-sided [0.691 to 1.218]
Statistical Analysis 3: Comparison: Dabigatran vs Rivaroxaban (Dabigatran) vs Dabigatran vs Rivaroxaban (Rivaroxaban); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.771, 95% CI 2-sided [0.578 to 1.027]

15. Secondary Outcome: Event Rate of Other Bleeding Requiring Hospitalization: NOAC Versus Warfarin Analysis
Description: Event rate was defined as number of events divided by 100 participant-years for first occurrence of other bleeding events after index date was reported. Other bleeding requiring hospitalization was identified using hospital claims which had other bleeding KCD code (D62, H448, H3572, H356, H313, H210, H113, H052, H470, H431, I312, N020-N029, N421, N831, N857, N920, N923, N930, N938, N939, M250, R233, R040, R041, R042, R048, R049, T792, T810, N950, R310, R311, R318, R58, T455, Y442, D683). Index date = the first prescription date of study drugs during intake duration. Participants were identified as NOAC user or Warfarin user depending on the date when they first used NOAC or Warfarin during intake duration.
Time Frame: Maximum of 1 year 4 months (From 1-July-2015 to 30-November-2016)
Population: as for outcome 1
Measure: Number; unit: events per 100 participants-years
Arm/Group | Apixaban vs Warfarin (Apixaban) | Apixaban vs Warfarin (Warfarin) | Dabigatran vs Warfarin (Dabigatran) | Dabigatran vs Warfarin (Warfarin) | Rivaroxaban vs Warfarin (Rivaroxaban) | Rivaroxaban vs Warfarin (Warfarin)
Number analyzed (Participants) | 10514 | 8677 | 11415 | 8676 | 17780 | 8638
events per 100 participants-years | 3.75 | 6.93 | 3.86 | 6.61 | 4.42 | 6.85
Statistical Analysis 1: Comparison: Apixaban vs Warfarin (Apixaban) vs Apixaban vs Warfarin (Warfarin); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.581, 95% CI 2-sided [0.481 to 0.701]
Statistical Analysis 2: Comparison: Dabigatran vs Warfarin (Dabigatran) vs Dabigatran vs Warfarin (Warfarin); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.640, 95% CI 2-sided [0.534 to 0.766]
Statistical Analysis 3: Comparison: Rivaroxaban vs Warfarin (Rivaroxaban) vs Rivaroxaban vs Warfarin (Warfarin); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.838, 95% CI 2-sided [0.622 to 1.130] — HR evaluated using extended Cox model

16. Secondary Outcome: Event Rate of Other Bleeding Requiring Hospitalization: NOAC Versus NOAC Analysis
Description: Event rate was defined as number of events divided by 100 participant-years for first occurrence of other bleeding events after index date was reported. Other bleeding requiring hospitalization was identified using hospital claims which had other bleeding KCD code (D62, H448, H3572, H356, H313, H210, H113, H052, H470, H431, I312, N020-N029, N421, N831, N857, N920, N923, N930, N938, N939, M250, R233, R040, R041, R042, R048, R049, T792, T810, N950, R310, R311, R318, R58, T455, Y442, D683). Index date = the first prescription date of study drugs during intake duration.
Time Frame: Maximum of 1 year 4 months (From 1-July-2015 to 30-November-2016)
Population: as for outcome 1
Measure: Number; unit: events per 100 participants-years
Arm/Group | Apixaban vs Dabigatran (Apixaban) | Apixaban vs Dabigatran (Dabigatran) | Apixaban vs Rivaroxaban (Apixaban) | Apixaban vs Rivaroxaban (Rivaroxaban) | Dabigatran vs Rivaroxaban (Dabigatran) | Dabigatran vs Rivaroxaban (Rivaroxaban)
Number analyzed (Participants) | 10514 | 11415 | 10514 | 17780 | 11415 | 17779
events per 100 participants-years | 3.67 | 4.06 | 3.73 | 4.54 | 3.83 | 4.35
Statistical Analysis 1: Comparison: Apixaban vs Dabigatran (Apixaban) vs Apixaban vs Dabigatran (Dabigatran); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.881, 95% CI 2-sided [0.732 to 1.061]
Statistical Analysis 2: Comparison: Apixaban vs Rivaroxaban (Apixaban) vs Apixaban vs Rivaroxaban (Rivaroxaban); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.802, 95% CI 2-sided [0.678 to 0.947]
Statistical Analysis 3: Comparison: Dabigatran vs Rivaroxaban (Dabigatran) vs Dabigatran vs Rivaroxaban (Rivaroxaban); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Hazard Ratio (HR) = 0.882, 95% CI 2-sided [0.754 to 1.032]

ADVERSE EVENTS:
Time Frame: Not applicable as safety data was not planned to be collected during the study
Description: Safety data was not planned to be collected during the study.
Arm/Group | NOAC - Apixaban | NOAC - Dabigatran | NOAC - Rivaroxaban | Warfarin | Aspirin
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Data for Aspirin group could not be matched with other treatment groups (because of genuine difference and heterogeneity in their characteristics) using IPTW method. Hence, no data for Aspirin reporting arm is reported in outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-05-03): https://cdn.clinicaltrials.gov/large-docs/72/NCT03572972/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-03): https://cdn.clinicaltrials.gov/large-docs/72/NCT03572972/SAP_001.pdf